CLINICAL TRIAL: NCT07299578
Title: A Study of Sleep Disorders and Their Impact on Patients With Ménière's Disease
Brief Title: Sleep Disorders and Their Impact on Patients With Ménière's Disease
Acronym: SoM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9380
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sleep Disorders
Keywords: Sleep Disorder; Ménière's Disease
MeSH Terms: conditions — Sleep Wake Disorders; Meniere Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ménière's disease was first described by Prosper Ménière in 1861 as a balance disorder originating in the inner ear. It is diagnosed based on a characteristic clinical triad of low-frequency hearing loss, tinnitus, and vertigo attacks. The underlying cause is thought to be a pressure imbalance in the inner ear between the endolymphatic and perilymphatic sectors.

The prevalence of Ménière's disease ranges from 34 to 190 per 100,000 inhabitants.

The physiology of Ménière's disease is not yet fully understood. It appears that sleep disorders may be related.

In its 2016 report on Ménière's disease, the French Society of Otolaryngology (SÖL) recommends sleep studies for patients with Ménière's disease.

However, these recommendations are based on few studies, which is why we wanted to conduct this research.

The main hypothesis is the existence of a link between debilitating vertigo and sleep disturbances in patients with Ménière's disease.

In cases of more significant sleep disturbances in patients with debilitating Ménière's disease, it is important to focus more thoroughly on these disturbances during ENT consultations, which are an integral part of effective multidisciplinary care.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Patient followed for Ménière's disease in the ENT department at Strasbourg University Hospital between June 1, 2019, and January 31, 2021.

Exclusion Criteria:

* History of intracranial surgery or degenerative neurological disease.
* No prior sleep medicine consultations.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) followed for Ménière's disease in the ENT department at Strasbourg University Hospital between June 1, 2019, and January 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Vertigo-related disability Score AAO-HNS | 1 hour after consultation
  * Vertigo-related disability score AAO-HNS (American Academy of Otolaryngology-Head and Neck Surgery Functional Scale)
  * Vertigo is considered debilitating if the score is greater than 3 out of 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France